CLINICAL TRIAL: NCT03934528
Title: The Impact of Simulated Arm Movement Within a Virtual Reality Environment on Phantom Limb Pain in Upper Limb Amputees: A Pilot Study
Brief Title: The Impact of a Virtual Reality Environment on Phantom Limb Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to proceed during lockdown; post-lockdown vendor no longer supports the hardware on which the study was developed
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Stephen Pettifer, Professor, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS:259344
Record Dates: First submitted 2019-04-23; First posted 2019-05-02 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Phantom Limb Syndrome With Pain
Keywords: Phantom Limb Pain; Virtual Reality; Virtual Environment
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Study (Experimental)
  Interventions: Device: Virtual environment activity

INTERVENTIONS:
Device: Virtual environment activity — Patients undertake an activity using simulated arm movement within a virtual reality environment every day for two months

SUMMARY:
Phantom limb pain occurs in the majority of people who lose a limb. It significantly affects quality of life and is hard to manage. Recent evidence suggests that mirror therapy and similar techniques that create a visual representation of the missing limb under the control of the patient may reduce phantom limb pain.

The investigators previously explored the use of a virtual reality environment for this purpose with people with upper limb loss but found that using it within the clinical setting limited its potential efficacy. Phantom limb pain is highly variable and assessing the effects of the activity during a hospital appointment when the phantom pain may not be present, or may not be problematic, made it difficult to judge the effects adequately.

This study involves training the patient in the clinic to use a portable, self-contained virtual reality system which they will then use at home, unsupervised, for 2 months. The aim is to discover whether phantom limb pain intensity decreases by performing an activity in a virtual reality environment in which a visual representation of the missing limb is controlled by the patient. Participants will be directed to use the system every day, and whenever their phantom limb pain is present and problematic.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Unilateral upper limb amputee (transradial and transhumeral).
* Amputation occurred at least 6 months ago.
* Stump has fully healed and has no ulcerations present.

Exclusion Criteria:

* Amputation of digit(s) only.
* The presence of a wound, ulcer or broken skin on the residual limb.
* The presence of a psychiatric disorder.
* Have pre-existing binocular vision abnormalities.
* A history of seizures or epilepsy.
* A pacemaker or other implanted medical device that could be affected by magnets or components that emit radio waves.
* Lacking the capacity to understand the instructions on how to use the virtual reality equipment.
* Lacking the capacity to consent.
* Unable to comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in intensity of phantom limb pain using a numerical rating scale: 0=no pain present to 10=worst imaginable pain. | 2 months

SECONDARY OUTCOMES:
Change from baseline of number of phantom limb pain episodes per month. | 2 months
Change from baseline of average duration of phantom limb pain episodes. | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom